CLINICAL TRIAL: NCT05570149
Title: EptinezuMaB in ReAl-world evidenCE: a 12-Months, Multicenter, Real-Life, Cohort Study in High-Frequency Episodic and Chronic Migraine (the EMBRACE Study)
Brief Title: EptinezuMaB in ReAl-world evidenCE: Multicenter, Real Life, Cohort Study in Migraine.
Acronym: EMBRACE
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 177/SR/24
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Migraine Disorders
Keywords: Eptinezumab,; Calcitonin gene-related peptide,; Effectiveness,; Real-life,; Migraine,; Safety; Treatment
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab; Saline Solution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Eptinezumab 100 mg or Eptinezumab 300 mg administered intravenously in 100 mL saline solution — migraine prophylaxis
  Other Names: anti CGRP monoclonal antibody

SUMMARY:
The object of this study is to assess the effectiveness, safety, and tolerability of eptinezumab in a real life migraine population.

DETAILED DESCRIPTION:
Eptinezumab is an humanized IgG1 and the only antiCGRP mAb administered intravenously by a quarterly dosing regimen. In randomized-controlled studies (RCTs), eptinezumab proved to be effective in preventing episodic and chronic migraine even in patients with 2 to 4 prior preventive failures and in shortening the time to complete migraine freedom when infused during a moderate-to severe migraine attack. Eptinezumab 100 mg can be used for the first administration and later if deemed necessary, the dose upgraded to 300 mg.

EMBRACE is a multicenter, prospective, cohort, real-life study carried out in Italian headache centers. Consecutive patients with high frequency episodic (HFEM: ≥8 migraine days/month) or CM (≥15 headache days/month), according to The International Classification of Headache Disorders, 3rd edition (ICHD-III), referred to participating centers. The aim of this study is to assess effectiveness, safety and tolerability of eptinezumab 100 mg iv or 300 mg iv with a quarterly dosing regimen in a real-world migraine patients population.

ELIGIBILITY:
KEY INCLUSION CRITERIA

1. Age between 18 and 75 years;
2. Males and females;
3. Willingness to sign the informed consent;
4. High frequency episodic migraine, at least 8 days per month of disabling migraine in the past 3 months;
5. Chronic migraine, according to the ICHD-III criteria;

KEY EXCLUSION CRITERIA

1. Other headaches different than migraine;
2. Known intolerance to eptinezumab or eccipients;
3. Current treatment with other mAbs;
4. Vascular disease or Raynaud.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients aged 18-75 affected by hight frequency or chronic migraine with or without medication overuse.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in monthly migraine days (MMD) in HFEM or monthly headache days (MHD) in CM; | over 12 weeks of treatment compared to baseline
  assessment of MMD or MHD
Change from baseline in MMD in HFEM or MHD in CM; | over 24 weeks of treatment compared to baseline
  assessment of MMD or MHD
Change from baseline in MMD in HFEM or MHD in CM; | over 48 weeks of treatment compared to baseline
  assessment of MMD or MHD
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | over 12 months of treatment compared to baseline
  assessment of occurrence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Change in monthly analgesic intake | over 12 weeks compared to baseline
  Assessment of monthly analgesic intake
Change in monthly analgesic intake | over 24 weeks compared to baseline
  Assessment of monthly analgesic intake
Change in monthly analgesic intake | over 48 weeks compared to baseline
  Assessment of monthly analgesic intake
Change in Numeric Rating Scale (NRS) | over 12 weeks compared to baseline
  Assessment of NRS
Change in Numeric Rating Scale (NRS) | over 24 weeks compared to baseline
  Assessment of NRS
Change in Numeric Rating Scale (NRS) | over 48 weeks compared to baseline
  Assessment of NRS
Change in Headache Impact Test-6 (HIT-6) | over 12 weeks compared to baseline
  Assessment of HIT-6
Change in Headache Impact Test-6 (HIT-6) | over 24 weeks compared to baseline
  Assessment of HIT-6
Change in Headache Impact Test-6 (HIT-6) | over 48 weeks compared to baseline
  Assessment of HIT-6
Change in Migraine Disability Assessment Score (MIDAS) | over 12 weeks compared to baseline
  Assessment of MIDAS
Change in Migraine Disability Assessment Score (MIDAS) | over 24 weeks compared to baseline
  Assessment of MIDAS
Change in Migraine Disability Assessment Score (MIDAS) | over 48 weeks compared to baseline
  Assessment of MIDAS
Change in Migraine interictal burden (MIBS-4) | over 12 weeks compared to baseline
  Assessment of MIBS-4
Change in Migraine interictal burden (MIBS-4) | over 24 weeks compared to baseline
  Assessment of MIBS-4
Change in Migraine interictal burden (MIBS-4) | over 48 weeks compared to baseline
  Assessment of MIBS
Change in Patient Global Impression of change (PGIC) scale | over 12 weeks compared to baseline
  Assessment of MIBS
Change in Patient Global Impression of change (PGIC) scale | over 24 weeks compared to baseline
  Assessment of MIBS
Change in Patient Global Impression of change (PGIC) scale | over 48 weeks compared to baseline
  Assessment of MIBS
≥50%, ≥75% and 100% response rates | over 12 weeks compared to baseline
  Assessment of responder rates
≥50%, ≥75% and 100% response rates | over 24 weeks compared to baseline
  Assessment of responder rates
≥50%, ≥75% and 100% response rates | over 48 weeks compared to baseline
  Assessment of responder rates
Percentage of migraine free patients on the day after dosing (infusion of eptinezumab) | the day after infusion of eptinezumab (first infusion of eptinezumab)
  Assessment of percentage of migraine free patients on the day after dosing (first infusion of eptinezumab)
Percentage of migraine free patients on the day after dosing (infusion of eptinezumab) | the day after infusion of eptinezumab (second infusion of eptinezumab)
  Assessment of percentage of migraine free patients on the day after dosing (second infusion of eptinezumab)
Proportion of patients with medication overuse at baseline reverting to no medication overuse | over 12 weeks compared to baseline
  Assessment of proportion of patients with medication overuse at baseline reverting to no medication overuse
Proportion of patients with medication overuse at baseline reverting to no medication overuse | over 24 weeks compared to baseline
  Assessment of proportion of patients with medication overuse at baseline reverting to no medication overuse
Proportion of patients with medication overuse at baseline reverting to no medication overuse | over 48 weeks compared to baseline
  Assessment of proportion of patients with medication overuse at baseline reverting to no medication overuse

CONTACTS AND LOCATIONS:
Overall Officials: Piero Barbanti, MD, PhD, Study Chair — IRCCS San Raffaele Roma
Locations (1):
- IRCCS San Raffaele Roma, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashina M, Saper J, Cady R, Schaeffler BA, Biondi DM, Hirman J, Pederson S, Allan B, Smith J. Eptinezumab in episodic migraine: A randomized, double-blind, placebo-controlled study (PROMISE-1). Cephalalgia. 2020 Mar;40(3):241-254. doi: 10.1177/0333102420905132. Epub 2020 Feb 19. PMID 32075406
- [Background] Villar-Martinez MD, Moreno-Ajona D, Goadsby PJ. Eptinezumab for the preventive treatment of migraine. Pain Manag. 2021 Mar;11(2):113-121. doi: 10.2217/pmt-2020-0075. Epub 2020 Dec 7. PMID 33280422
- [Background] Lipton RB, Goadsby PJ, Smith J, Schaeffler BA, Biondi DM, Hirman J, Pederson S, Allan B, Cady R. Efficacy and safety of eptinezumab in patients with chronic migraine: PROMISE-2. Neurology. 2020 Mar 31;94(13):e1365-e1377. doi: 10.1212/WNL.0000000000009169. Epub 2020 Mar 24. PMID 32209650
- [Background] Ashina M, Lanteri-Minet M, Pozo-Rosich P, Ettrup A, Christoffersen CL, Josiassen MK, Phul R, Sperling B. Safety and efficacy of eptinezumab for migraine prevention in patients with two-to-four previous preventive treatment failures (DELIVER): a multi-arm, randomised, double-blind, placebo-controlled, phase 3b trial. Lancet Neurol. 2022 Jul;21(7):597-607. doi: 10.1016/S1474-4422(22)00185-5. PMID 35716692